CLINICAL TRIAL: NCT03992495
Title: The Effect of Exercise on Neck Pain and Pain Sensitivity
Brief Title: The Effect of Exercise on Pain Sensitivity in a Population With Ongoing Neck Pain Compared to Healthy Controls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Steffan Wittrup Christensen, Assistant professor, Aalborg University
Other Study IDs: N-20180063_Sub-project_3
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Neck Pain; Healthy
Keywords: Exercise; Neck pain; Pain sensitivity
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neck pain: People suffering from neck pain at the time of recruitment
  Interventions: Other: Exercise
- Healthy: Participants with no significant past neck pain, chronic pain or other relevant medical disorders.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — All participants will be exposed to aerobic/strengthening exercises

SUMMARY:
This study investigates the effect of exercise on pain sensitivity in ongoing neck pain patients compared to a healthy control group.

DETAILED DESCRIPTION:
Increased pain sensitivity is a common finding in neck pain patients when compared to healthy controls. Although most studies favor exercise as an intervention, the specific effect on pain sensitivity is still debated. This study will investigate the effect of exercise on pain sensitivity in neck pain patients compared to healthy controls

ELIGIBILITY:
Inclusion Criteria: - Healthy participants

* Pain free healthy participants
* Able to speak, read and understand Danish and English

Exclusion Criteria: - Healthy participants

* Pain from the neck or shoulder area during the past 6 months
* Experience of delayed onset muscle soreness (DOMS) during the week leading up to the test session
* Former surgery in neck or shoulder
* Current or previous chronic or recurrent pain condition
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Regular use of analgesics
* Abnormally disrupted sleep in the last 24 hours preceding the experiment
* Lack of ability to cooperate

Inclusion Criteria: - Neck pain population

* Self reported neck pain lasting three months or longer.
* Able to speak, read and understand Danish and English
* Reduced/painful active range of motion of the head and/or painful reaction to palpation of the neck at the time of inclusion

Exclusion Criteria: - Neck pain population

* Shoulder pain during arm movements
* Experience of DOMS during the week leading up to the test session
* Former surgery in neck or shoulder
* Current or previous chronic or recurrent pain condition other than neck pain
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Abnormally disrupted sleep in the 24 hours preceding the experiment
* Lack of ability to cooperate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People with self-reported pain from the neck area with a symptom duration of three months or longer and pain free healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain sensitivity | Baseline, 6 weeks, 12 weeks
  Pain sensitivity will be estimated by determining the pressure pain threshold (PPT) on the neck before and after exercise

SECONDARY OUTCOMES:
Change in perceived pain | Baseline, 6 weeks, 12 weeks
  Pain will be scored using a scale from 0-10 with 0 being no pain and 10 being worst imaginable pain and by drawing perceived painful areas on a body charts
Change in disability | Baseline, 6 weeks, 12 weeks
  Disability will be estimated by scoring the Neck Disability Index (NDI) questionnaire. The questionnaire is designed to help express how neck pain affects your ability to manage everyday activities.(Domains: pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, recreation). Higher score = high level of disability

OTHER OUTCOMES:
Change in body movements | Baseline, 6 weeks, 12 weeks
  Head repositioning accuracy will be tested using a clinical test in a seated position. Participants will turn their head to end of range in from a neutral position with their eyes closed and return to the start position again. The difference between start and end position will be recorded. Standing balance will be assessed by recording the time (seconds) a tandem stance can be maintained.

CONTACTS AND LOCATIONS:
Overall Officials: Steffan W Christensen, PhD, Principal Investigator — Aalborg University

IPD SHARING:
Plan to Share IPD: Undecided